CLINICAL TRIAL: NCT03393754
Title: A Phase 3 Double-Blind Randomized Controlled Trial to Compare the Immunogenicity and Safety of a Three-dose Regimen of Sci-B-Vac® to a Three-dose Regimen of Engerix-B® in Adults (PROTECT)
Brief Title: Immunogenicity and Safety of Sci-B-Vac® to Engerix-B® in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VBI Vaccines Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Sci-B-Vac-001; 2017-001819-36 (EudraCT Number)
Record Dates: First submitted 2017-11-23; First posted 2018-01-08 (Actual); Results first posted 2020-07-07 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Hepatitis B Vaccines
Keywords: Hepatitis B Vaccines
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sci-B-Vac® Hepatitis B Vaccination (Experimental): Sci-B-Vac® (hepatitis B vaccine) Hepatitis B Vaccination, Solution, 10ug, IM injection at Days 0, 28, and 168.
  Interventions: Biological: Hepatitis B Vaccination
- Engerix-B® Hepatitis B Vaccination (Active Comparator): Engerix-B® (hepatitis B vaccine) Hepatitis B Vaccination, Solution, 20ug, IM injection at Days 0, 28, and 168.
  Interventions: Biological: Hepatitis B Vaccination

INTERVENTIONS:
Biological: Hepatitis B Vaccination — Prophylactic Hepatitis B Vaccination

SUMMARY:
This study is a double-blind randomized controlled trial designed to establish the non-inferiority of Sci-B-Vac® compared to Engerix-B® in adults ≥ 18 years old and the superiority of Sci-B-Vac® compared to Engerix-B® in ≥ 45 years old.

DETAILED DESCRIPTION:
This study is a double-blind randomized controlled trial designed to establish the non-inferiority of Sci-B-Vac® compared to Engerix-B® in adults ≥ 18 years old and the superiority of Sci-B-Vac® compared to Engerix-B® in adults ≥ 45 years old. Study subjects are randomized 1:1 to receive either a total of 3 injections of Sci-B-Vac® or 3 injections of Engerix-B® intra-muscularly (IM) on Days 0, 28, and 168.

ELIGIBILITY:
Inclusion Criteria:

* Any gender.
* Age ≥ 18 years
* In stable health as determined by a physical examination and laboratory tests values. Common chronic conditions such as, but not limited to, type 2 diabetes, high blood pressure, Chronic Obstructive Pulmonary Disease (COPD) and asthma will be accepted if the condition is well controlled, as determined by the investigator, and not meeting the exclusion criteria. For subjects > 65 years old, Frailty Index ≤3
* If female, either is not of childbearing potential or is of childbearing potential and must agree to use an adequate birth control method during the screening period and until the end of her participation in the study
* Able and willing to give consent.

Exclusion Criteria:

* Previous vaccination with any Hep B vaccine (licensed or experimental).
* Treatment by immunosuppressant within 30 days of enrollment including but not limited to corticosteroids at a dose that is higher than an oral or injected physiological dose, or a prednisolone-equivalent dose > 20 mg /day (Inhaled and topical steroids are allowed).
* Known history of immunological function impairment
* Pregnancy or breastfeeding
* Immunization with attenuated vaccines (e.g. MMR) within 4 weeks prior to enrollment
* Immunization with inactivated vaccines (e.g. influenza) within 2 weeks prior to enrolment
* Has received blood products or immunoglobulin within 90 days of enrollment or is likely to require blood products during the study period
* Subject in another clinical trial with an investigational drug or a biologic within 30 days of enrollment
* Has received granulocyte-macrophage colony stimulating factor (G/GM-CSF) or erythropoietin (EPO) within 30 days of enrollment or likely to require GM-CSF or erythropoietin during the study period
* Any history of cancer requiring chemotherapy or radiation within 5 years of randomization or current disease.
* Any skin abnormality or tattoo that would limit post-vaccination injection site assessment
* History of allergic reactions or anaphylactic reaction to any vaccine component (Engerix-B® or Sci-B-Vac®)
* Unwilling, or unable in the opinion of the investigator, to comply with study requirements, including the use of an adequate birth control method
* Immediate family members of study center staff (parents, sibling, children)
* Current or past hepatitis B infection or prior vaccination as evidenced by HBV markers at screening
* Known hepatitis C infection or positive Hepatitis C serology at screening, unless treated and cured
* Known human immunodeficiency virus (HIV) infection or positive HIV serology at screening
* Renal impairment at screening
* Uncontrolled diabetes mellitus
* Uncontrolled hypertension
* Any laboratory test abnormality that would be considered of Grade 1 severity and is considered as clinically significant by the investigator. Grade 3 severity or above is exclusionary, regardless of clinical assessment.
* Diagnosis of advanced stage heart failure or Unstable Angina.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1607 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2019-04-08 (Actual); Study Completion 2019-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Diaz-Mitoma, MD, PhD, Study Director — VBI Vaccines
Locations (28):
- United States (10):
  - Accel Research Sites, Birmingham, Alabama
  - Anaheim Clinical Trials, Anaheim, California
  - Avail Clinical Research, DeLand, Florida
  - Suncoast Research Group, Miami, Florida
  - Clinical Research Atlanta, Atlanta, Georgia
  - Advanced Clinical Research, Boise, Idaho
  - Clinical Research Center of Nevada, Las Vegas, Nevada
  - Rapid Medical Research, Cleveland, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Advanced Clinical Research, Salt Lake City, Utah
- Universitair Ziekenhuis Gent, Ghent, Oost-Vlaanderen, Belgium
- Canada (7):
  - BC Children's Hospital Research Institute, Vancouver, British Columbia
  - University of Manitoba, Winnipeg, Manitoba
  - Canadian Center for Vaccinology, Halifax, Nova Scotia
  - Medicore Research Inc, Greater Sudbury, Ontario
  - Ottawa Hospital, Ottawa, Ontario
  - McGill University Health Centre, Montreal, Quebec
  - CHU de Québec Université Laval, Québec, Quebec
- Finland (10):
  - Espoo Vaccine Research Clinic, Espoo
  - Helsinki South Vaccine Research Clinic, Helsinki
  - Järvenpää Vaccine Research Clinic, Jarvenpaa
  - Kokkola Vaccine Research Clinic, Kokkola
  - Oulu Vaccine Research Clinic, Oulu
  - Pori Vaccine Research Clinic, Pori
  - Seinäjoki Vaccine Research Clinic, Seinäjoki
  - Tampere Vaccine Research Clinic, Tampere
  - University of Tampere, Tampere
  - Turku Vaccine Research Clinic, Turku

REFERENCES:
- [Derived] Berthoud TK, Ahmed T, Nadia W, Petrov I, Yang L, Colledge D, Hammond R, Soare C, Ontsouka B, Plaskin D, Anderson DE, Diaz-Mitoma F. A three antigen hepatitis B vaccine induces T cells to Pres1 and Pres2 which correlate with anti HBs antibody titers: An investigation into the immunological mechanisms contributing to high anti-HBs titers. Vaccine. 2025 Jan 1;43(Pt 2):126513. doi: 10.1016/j.vaccine.2024.126513. Epub 2024 Nov 12. PMID 39536477
- [Derived] Talbird SE, Anderson SA, Nossov M, Beattie N, Rak AT, Diaz-Mitoma F. Cost-effectiveness of a 3-antigen versus single-antigen vaccine for the prevention of hepatitis B in adults in the United States. Vaccine. 2023 May 26;41(23):3506-3517. doi: 10.1016/j.vaccine.2023.04.022. Epub 2023 May 3. PMID 37147201
- [Derived] Vesikari T, Langley JM, Segall N, Ward BJ, Cooper C, Poliquin G, Smith B, Gantt S, McElhaney JE, Dionne M, van Damme P, Leroux-Roels I, Leroux-Roels G, Machluf N, Spaans JN, Yassin-Rajkumar B, Anderson DE, Popovic V, Diaz-Mitoma F; PROTECT Study Group. Immunogenicity and safety of a tri-antigenic versus a mono-antigenic hepatitis B vaccine in adults (PROTECT): a randomised, double-blind, phase 3 trial. Lancet Infect Dis. 2021 Sep;21(9):1271-1281. doi: 10.1016/S1473-3099(20)30780-5. Epub 2021 May 11. PMID 33989539

RESULTS

PARTICIPANT FLOW:
Groups:
- Engerix-B® Hepatitis B Vaccination: Engerix-B® (hepatitis B vaccine) Hepatitis B Vaccination, Solution, 20ug, intramuscular (IM) injection at Days 0, 28, and 168.
  Hepatitis B Vaccination: Prophylactic Hepatitis B Vaccination
- Sci-B-Vac® Hepatitis B Vaccination: Sci-B-Vac® (hepatitis B vaccine) Hepatitis B Vaccination, Solution, 10ug, intramuscular (IM) injection at Days 0, 28, and 168.
  Hepatitis B Vaccination: Prophylactic Hepatitis B Vaccination
Period: Overall Study
Arm/Group | Engerix-B® Hepatitis B Vaccination | Sci-B-Vac® Hepatitis B Vaccination
Started | 811 | 796
Completed | 785 | 758
Not Completed | 26 | 38

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Engerix-B® Hepatitis B Vaccination | Sci-B-Vac® Hepatitis B Vaccination | Total
Number analyzed (Participants) | 811 | 796 | 1607
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (13.46) | 56.6 (13.2) | 56.6 (58.0)
Age, Customized [Count of Participants; unit: Participants]
  18-44 years | 154 | 145 | 299
  45-64 years | 361 | 355 | 716
  ≥ 65 years | 296 | 296 | 592
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 508 | 481 | 989
  Male | 303 | 315 | 618
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 75 | 79 | 154
  Not Hispanic or Latino | 732 | 714 | 1446
  Unknown or Not Reported | 4 | 3 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 730 | 715 | 1445
  Asian | 4 | 8 | 12
  Black or African American | 65 | 66 | 131
  American Indian or Alaska Native | 4 | 5 | 9
  Native Hawaiian or other Pacific Islander | 0 | 1 | 1
  Other | 8 | 1 | 9
Region of Enrollment [Number; unit: participants]
  Canada | 133 | 126 | 259
  Europe | 336 | 332 | 668
  United States | 342 | 338 | 680
BMI category [Count of Participants; unit: Participants]
  >30 kg/m^2 | 292 | 297 | 589
  <=30 kg/m^2 | 519 | 499 | 1018
Smoking status/Tobacco use [Count of Participants; unit: Participants]
  Current smoker/tobacco user | 113 | 104 | 217
  Former smoker/tobacco user | 224 | 203 | 427
  Non-smoker/non-tobacco user | 474 | 489 | 963
Diabetes status [Count of Participants; unit: Participants]
  Diabetic | 65 | 60 | 125
  Non-diabetic | 746 | 736 | 1482

OUTCOME MEASURES:

1. Primary Outcome: Seroprotection Rate (SPR) Defined as Percentage of Adults ≥ 18 Years Old Achieving Anti-HBs Levels of ≥10 mIU/mL in Serum at Study Day 196
Description: To demonstrate that the SPR 4 weeks after completion of the three-dose regimen of Sci-B-Vac® is non-inferior to a three-dose regimen of Engerix-B® in adults ≥18 years old; i.e. the lower bound of the 95% two-sided confidence interval (CI) of the difference between the SPR in the Sci-B-Vac® arm minus the SPR in the Engerix-B® arm, achieved 4 weeks after the third vaccination, will be > - 5%.
Time Frame: Day 196
Population: Per-protocol set - all subjects in the full analysis set who received all 3 injections, had at least baseline and 1 post-baseline immunogenicity assessment (at the time point of interest), were seronegative at baseline, and had no major protocol deviations leading to exclusion.
Measure: Number (95% Confidence Interval); unit: percentage of participants seroprotected
Arm/Group | Engerix-B® Hepatitis B Vaccination | Sci-B-Vac® Hepatitis B Vaccination
Number analyzed (Participants) | 723 | 718
percentage of participants seroprotected | 76.49 [73.22 to 79.53] | 91.36 [89.07 to 93.32]

2. Primary Outcome: Seroprotection Rate (SPR) Defined as Percentage of Adults ≥ 45 Years Old Achieving Anti-HBs Levels of ≥10 mIU/mL in Serum at Study Day 196
Description: To demonstrate that the SPR 4 weeks after completion of the three-dose regimen of Sci-B-Vac® is superior to the SPR 4 weeks after completion of the three-dose regimen of Engerix-B® in older adults ≥ 45 years old i.e. the lower bound of the 95% two-sided CI of the difference between the SPR in the Sci-B-Vac® arm minus the SPR in the Engerix-B® arm, achieved 4 weeks after receiving the third vaccination, will be > 5%.
Time Frame: Day 196
Population: Full analysis set - subjects who received at least 1 injection and had at least baseline and 1 post baseline immunogenicity assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants seroprotected
Arm/Group | Engerix-B® Hepatitis B Vaccination | Sci-B-Vac® Hepatitis B Vaccination
Number analyzed (Participants) | 627 | 625
percentage of participants seroprotected | 73.05 [69.39 to 76.48] | 89.44 [86.76 to 91.74]

3. Secondary Outcome: Percentage of Subject-reporting Solicited Local and Systemic Adverse Events (AEs)
Description: Analysis of local and systemic solicited adverse events with an interval of onset of Day 1 to Day 7 after any vaccination with either Sci-B-Vac® or Engerix-B®, in adults ≥18 years old.
Time Frame: Day of vaccine administration and six subsequent days
Population: Safety set: all subjects in the All Enrolled Set who received at least 1 injection
Measure: Count of Participants; unit: Participants
Arm/Group | Engerix-B® Hepatitis B Vaccination | Sci-B-Vac® Hepatitis B Vaccination
Number analyzed (Participants) | 811 | 796
Participants
  Pain | 294 | 503
  Tenderness | 282 | 484
  Pruritus/itching | 66 | 76
  Redness/erythema | 15 | 18
  Swelling/edema | 12 | 18
  Fatigue | 249 | 242
  Headache | 238 | 249
  Myalgia | 197 | 276
  Diarrhea | 96 | 82
  Nausea/vomiting | 73 | 56

ADVERSE EVENTS:
Time Frame: 1 year
Description: Number (%) of subject-reporting unsolicited adverse events (AEs) and serious adverse events (SAEs).
Arm/Group | Engerix-B® Hepatitis B Vaccination | Sci-B-Vac® Hepatitis B Vaccination
All-Cause Mortality (participants affected / at risk) | 0/811 | 0/796
Serious Adverse Events (participants affected / at risk) | 21/811 | 32/796
Other Adverse Events (participants affected / at risk) | 455/811 | 429/796
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Engerix-B® Hepatitis B Vaccination (N=811) | Sci-B-Vac® Hepatitis B Vaccination (N=796)
Atrial fibrillation (Cardiac disorders) | 2 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Nodal arrhythmia (Cardiac disorders) | 0 | 1
Trisomy 21 (Congenital, familial and genetic disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Diaphragmatic hernia (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 | 1
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Escherichia sepsis (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Gastrointestinal infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1
Back injury (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1
Troponin increased (Investigations) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Peroneal nerve palsy (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Subchorionic haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Aortic stenosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Engerix-B® Hepatitis B Vaccination (N=811) | Sci-B-Vac® Hepatitis B Vaccination (N=796)
Diarrhoea (Gastrointestinal disorders) | 21 | 12
Toothache (Gastrointestinal disorders) | 10 | 5
Nausea (Gastrointestinal disorders) | 10 | 3
Fatigue (General disorders) | 40 | 34
Injection site pain (General disorders) | 13 | 23
Upper respiratory tract infection (Infections and infestations) | 57 | 51
Nasopharyngitis (Infections and infestations) | 32 | 37
Urinary tract infection (Infections and infestations) | 17 | 18
Sinusitis (Infections and infestations) | 17 | 11
Gastroenteritis (Infections and infestations) | 7 | 11
Bronchitis (Infections and infestations) | 6 | 10
Influenza (Infections and infestations) | 10 | 6
Muscle strain (Injury, poisoning and procedural complications) | 6 | 9
Respiratory rate increased (Investigations) | 7 | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 34 | 30
Back pain (Musculoskeletal and connective tissue disorders) | 27 | 36
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 | 17
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16 | 13
Neck pain (Musculoskeletal and connective tissue disorders) | 10 | 8
Headache (Nervous system disorders) | 71 | 69
Dizziness (Nervous system disorders) | 11 | 12
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 18 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 9
Hypertension (Vascular disorders) | 13 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-07-17): https://cdn.clinicaltrials.gov/large-docs/54/NCT03393754/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-13): https://cdn.clinicaltrials.gov/large-docs/54/NCT03393754/SAP_001.pdf